CLINICAL TRIAL: NCT04676646
Title: Phase IV, Double-Blind, Placebo-Controlled, Randomized-Withdrawal Trial Evaluating Sodium Zirconium Cyclosilicate (SZC) for the Management of Hyperkalaemia in Patients With Symptomatic Heart Failure With Reduced Ejection Fraction and Receiving Spironolactone
Brief Title: Study to Assess Efficacy and Safety of SZC for the Management of High Potassium in Patients With Symptomatic HFrEF Receiving Spironolactone
Acronym: REALIZE-K
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9480C00018; 2020-003312-27 (EudraCT Number)
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hyperkalaemia; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; Spironolactone

STUDY DESIGN:
Intervention Model Description: REALIZE-K is a Phase 4, multinational, multicenter, double-blind, placebo-controlled, randomized-withdrawal, parallel-group study.
Who Masked: Participant, Investigator
Masking Description: All participants entering the double-blind, randomised treatment period will be centrally assigned to randomised study intervention using an Interactive Response Technology/Randomisation and Trial Supply Management (IRT/RTSM). Randomisation will be stratified by the sK+ cohort determined by central laboratory at the start of the open-label phase (Day 1). Before the study is initiated, the telephone number and call-in directions for the IRT and/or the log in information and directions for the RTSM will be provided to each site.
  The IRT/RTSM will provide to the investigator(s) or pharmacists the kit identification number to be allocated to the participant at the dispensing visit. Routines for this will be described in the IRT/RTSM user manual that will be provided to each centre.
  The randomisation code should not be broken except in medical emergencies when the appropriate management of the participant requires knowledge of the treatment randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-label run-in phase (Experimental): Cohort 1 (4 weeks duration): Patients who are hyperkalemic at study entry will begin SZC 10 g TID for up to 48 hours followed by SZC 10 g once daily to achieve and maintain normokalemia. The SZC dose will be adjusted as needed to maintain normokalemia (dose range = 5 g every other day, to 5-15 g once daily).
  Cohort 2 (up to 6 weeks duration): Patients who develop hyperkalemia during the uptitration of spironolactone will receive SZC 10 g TID for up to 48 hours followed by SZC 10 g once daily to achieve and maintain normokalemia. The SZC dose will be adjusted as needed to maintain normokalemia (dose range = 5 g every other day, to 5-15 g once daily).
  Interventions: Drug: Sodium zirconium cyclosilicate; Drug: Placebo; Other: Spironolactone
- Randomized withdrawal phase (6 months) (Experimental): SZC arm and Placebo arm: Patients will continue on the SZC dose they were receiving at the end of the run-in phase.
  The SZC / Placebo dose will be adjusted as needed to maintain normokalemia (dose range = 5 g every other day, to 5-15 g once daily).
  Interventions: Drug: Sodium zirconium cyclosilicate; Drug: Placebo; Other: Spironolactone

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — Investigational medicinal product
  Other Names: SZC
Drug: Placebo — Placebo comparator
Other: Spironolactone — Background intervention.
  During the run-in phase, spironolactone will be initiated/uptitrated up to a maximum of 50 mg per day. During the randomized withdrawal phase the spironolactone dose at the end of the run-in phase will be maintained.

SUMMARY:
The main objective of this study is to evaluate the efficacy of SZC as compared with placebo in keeping potassium levels within the normal range (3.5-5.0 mEq/L) while on spironolactone ≥25 mg daily without assistance of rescue therapy for hyperkalaemia (HK).

DETAILED DESCRIPTION:
REALIZE-K is a Phase 4, multinational, multicenter, double-blind, placebo-controlled, randomized-withdrawal, parallel-group study that includes the following 3 phases: screening, 4-6 week open-label run-in phase where sodium zirconium cyclosilicate (SZC) and spironolactone will be optimized, followed by a 6-month double-blind, placebo-controlled, randomized withdrawal treatment phase.

Patients meeting the following criteria will enter the 4-6 week open-label run-in phase: symptomatic heart failure with reduced ejection fraction (HFrEF); receiving an angiotensin-converting enzyme inhibitor (ACEi), angiotensin II receptor blocker (ARB), or angiotensin receptor-Neprilysin inhibitor (ARNi); receiving no spironolactone or eplerenone, or receiving low-dose spironolactone (<25 mg daily); receiving a beta-blocker unless contraindicated; AND with hyperkalemia (sK+ 5.1-5.9 mEq/L) and an eGFR >/= 30 mL/min/1.73m2, OR normokalemic (sK+ 3.5-5.0 mEq/L) and 'at risk' of developing hyperkalemia (ie, history of hyperkalemia within the past 36 months and eGFR >/= 30 mL/min/1.73m2, or sK+ 4.5-5.0 mEq/L and eGFR 30-60 mL/min/1.73m2 and/or age >75 years).

Patients who are normokalemic on SZC and receiving spironolactone >/= 25 mg daily at the end of the open-label run-in phase will enter the 6-month double-blind, placebo-controlled, randomized withdrawal treatment phase. Eligible patients will be randomized 1:1, stratified by run-in phase sK+ cohort.

ELIGIBILITY:
INCLUSION CRITERIA

* Adults aged ≥18 years
* Potassium and estimated glomerular filtration rate (eGFR):
* Cohort 1: sK+ 5.1-5.9 mEq/L at screening/study enrolment and eGFR ≥30 mL/min/1.73 m2; OR
* Cohort 2: Normokalaemic (sK+ 3.5-5.0 mEq/L) at screening and 'at risk' of developing HK defined as any of the following:
* Have a history of HK (sK+ >5.0 mEq/L) within the prior 36 months and eGFR ≥30 mL/min/1.73 m2; or
* sK+ 4.5-5.0 mEq/L and eGFR 30 to 60 mL/min/1.73 m2; or
* sK+ 4.5-5.0 mEq/L, and age >75 years
* Symptomatic HFrEF (New York Heart Association [NYHA] class II-IV), which has been present for at least 3 months
* Left ventricular ejection fraction (LVEF) ≤40%
* Receiving angiotensin-converting enzyme inhibitor (ACEi), angiotensin II receptor blocker (ARB), or angiotensin receptor-Neprilysin inhibitor (ARNi)
* Not on or on low-dose spironolactone or eplerenone (<25 mg daily)
* Receiving beta-blocker unless contraindicated

EXCLUSION CRITERIA

* Heart failure due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy, or severe stenotic valve disease as a primary cause of HF
* Current inpatient hospitalisation with unstable HF, defined as any of the following:
* Systolic blood pressure <95 mmHg during the 6 hours prior to screening.
* Intravenous diuretic therapy during the 12 hours prior to screening.
* Use of intravenous inotropic drugs during the 24 hours prior to screening.
* Received mechanical circulatory support during the 48 hours prior to screening
* Previous cardiac transplantation or implantation of a ventricular assistance device (VAD) or similar device, or transplantation or implantation expected after randomisation

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (12):
  - Research Site, Fairhope, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Torrance, California
  - Research Site, Evanston, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Falls Church, Virginia
- Brazil (13):
  - Research Site, Belo Horizonte
  - Research Site, Bragança Paulista
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Canoas
  - Research Site, Joinville
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, Santa Cruz do Sul
  - Research Site, São Paulo
  - Research Site, Votuporanga
- Canada (8):
  - Research Site, Cambridge, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Whitby, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Terrebonne, Quebec
- Czechia (7):
  - Research Site, Brandýs nad Labem
  - Research Site, Broumov
  - Research Site, Hradec Králové
  - Research Site, Jaroměř
  - Research Site, Louny
  - Research Site, Ostrava
  - Research Site, Uherské Hradiště
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Zalaegerszeg
- Poland (5):
  - Research Site, Gdynia
  - Research Site, Lodz
  - Research Site, Lódz
  - Research Site, Skórzewo
  - Research Site, Żarów
- Spain (19):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Jaén
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (9):
  - Research Site, Ashington
  - Research Site, Bridgend
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Newport
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kosiborod MN, Cherney DZI, Desai AS, Testani JM, Verma S, Chinnakondepalli K, Dolling D, Patel S, Dahl M, Eudicone JM, Friberg L, Ouwens M, Antunes MO, Connelly KA, Madrini V Jr, Kuthi L, Lala A, Lorenzo M, Guimaraes PO, Marcos MC, Merkely B, Nunez J, Squire I, Vaclavik J, Wranicz J, Petrie MC. Sodium Zirconium Cyclosilicate for Management of Hyperkalemia During Spironolactone Optimization in Patients With Heart Failure. J Am Coll Cardiol. 2025 Mar 18;85(10):971-984. doi: 10.1016/j.jacc.2024.11.014. Epub 2024 Nov 18. PMID 39566872
- [Derived] Kosiborod MN, Cherney D, Connelly K, Desai AS, Guimaraes PO, Kuthi L, Lala A, Madrini V Jr, Merkely B, Villota JN, Squire I, Testani JM, Vaclavik J, Verma S, Wranicz J, Dahl M, Eudicone JM, Friberg L, Petrie MC. Sodium Zirconium Cyclosilicate in HFrEF and Hyperkalemia: REALIZE-K Design and Baseline Characteristics. JACC Heart Fail. 2024 Oct;12(10):1707-1716. doi: 10.1016/j.jchf.2024.05.003. Epub 2024 May 13. PMID 38878009
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00018&attachmentIdentifier=e57bd34e-2d30-4052-8cac-bea3b1f3ab81&fileName=D9480C00018_Redacted_SAP.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00018&attachmentIdentifier=77d3fb06-6ea2-4c65-ae70-716e2640df90&fileName=D9480C00018_redacted_CSP.pdf&versionIdentifier=
- See also: redacted CSR study synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00018&attachmentIdentifier=16f75da0-06f2-4e73-ac6f-bb3b1a8310da&fileName=D9480C00018_redacted_CSR_study_synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of two phases, an open-label run-in phase and a placebo-controlled randomized-withdrawal phase.
  Of the 366 participants enrolled in the open-label run-in phase, 203 participants entered into the randomized-withdrawal phase (102 received SZC treatment and 101 received placebo).
Groups:
- Open-label Run-in Phase: Participants with symptomatic heart failure with reduced ejection fraction who were taking no or low-dose spironolactone or eplerenone (< 25 mg daily) at screening were enrolled and allocated to Cohort 1 (hyperkalaemic at study entry) or Cohort 2 (normokalaemic at study entry).
- Randomized-withdrawal Phase - SZC Group: Participants continued on the SZC and spironolactone dose they were receiving at the end of the run-in phase.
- Randomized-withdrawal Phase - Placebo Group: Participants continued on the placebo and spironolactone dose they were receiving at the end of the run-in phase.
Period: Open-label Run-in Phase
Arm/Group | Open-label Run-in Phase | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Started | 366 | 0 | 0
Completed | 203 | 0 | 0
Not Completed | 163 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Study-specific Withdrawal Criteria | 2 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 144 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Withdrawn from study due to withdrawal by co-investigator | 1 | 0 | 0
Not completed — Withdrawn from study due to withdrawal by PI | 1 | 0 | 0
Period: Randomised-withdrawal Phase
Arm/Group | Open-label Run-in Phase | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Started | 0 | 102 | 101
Completed | 0 | 88 | 87
Not Completed | 0 | 14 | 14
Not completed — Adverse Event | 0 | 5 | 5
Not completed — Death | 0 | 1 | 2
Not completed — Development of Study-specific Withdrawal Criteria | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawn from study due to PD - Wrong doses of spironolactone | 0 | 1 | 0
Not completed — Withdrawn from study due to spironolactone was stopped on May 28, related hyperkalaemia | 0 | 1 | 0
Not completed — Withdrawn from study due to the participant did not have enough medication by issues in IWRS | 0 | 0 | 1
Not completed — Withdrawn from study due to the patient was random by mistake on this date he was an OLRIF | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening
  Years | 72.5 (7.88) | 69.2 (10.46) | 70.9 (9.39)
Age, Customized [Number; unit: Participants]
  18-64 years | 18 | 32 | 50
  65-84 years | 79 | 63 | 142
  >=85 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 76 | 75 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 27 | 67
  Not Hispanic or Latino | 62 | 74 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 91 | 94 | 185
  Black or African American | 5 | 5 | 10
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 0 | 0
  Other | 6 | 2 | 8
  Not Reported | 0 | 0 | 0
Country [Number; unit: Participants]
  BRA | 31 | 19 | 50
  CAN | 7 | 16 | 23
  CZE | 3 | 13 | 16
  ESP | 33 | 26 | 59
  GBR | 9 | 4 | 13
  HUN | 5 | 5 | 10
  POL | 8 | 10 | 18
  USA | 6 | 8 | 14
Type 2 diabetes at baseline [Number; unit: Participants] — Coded using baseline medical history
  Participants
    Yes | 27 | 25 | 52
    No | 75 | 76 | 151

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved Response, Defined as Serum Potassium (sK+) Within 3.5 to 5.0 mEq/L, Spironolactone Greater Than or Equal to 25 mg Daily, no Rescue Therapy for Hyperkalaemia
Description: The median percentages of participants having a response are presented. Response means all three requirements were met. Non-response was indicated for participants lost to follow-up, including death.
  The treatment effect was analysed using a generalised estimating equation (GEE) model with a binomial family and a log link, a dependent variable of response per visit, fixed independent variables of randomised treatment, subject recruitment country, a per visit indicator variable and open-label period cohort. The common odds ratio was derived together with two-sided 95% confidence intervals.
Time Frame: From Month 1 (Visit 9) to Month 6 (Visit 14), up to 6 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 102 | 101
Percentage of participants | 72.1 | 35.7
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p < 0.001, GEE model; Odds Ratio (OR) = 4.45, 95% CI 2-sided [2.89 to 6.86] — An odds ratio greater than 1 indicated increased odds of response on SZC compared to placebo

2. Secondary Outcome: Participants Who Achieved Response, Defined as sK+ Within 3.5-5.0 mEq/L, on the Same Dose of Spironolactone as Randomisation, no Rescue Therapy for Hyperkalaemia
Description: The median percentages of participants who achieved a response are presented. Response means all three requirements were met. Non-response was indicated for participants lost to follow-up, including death.
  The analysis was performed using a GEE model with a binomial family and a log link, a dependent variable of response per visit, fixed independent variables of randomised treatment, subject recruitment country, a per visit indicator variable and open-label period cohort. The common odds ratio was derived together with two-sided 95% confidence intervals.
Time Frame: From Month 1 (Visit 9) to Month 6 (Visit 14), up to 6 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 102 | 101
Percentage of participants | 58.2 | 22.9
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p < 0.001, GEE model; Odds Ratio (OR) = 4.58, 95% CI 2-sided [2.78 to 7.55] — An odds ratio >1 indicated increased odds of response on SZC compared to placebo

3. Secondary Outcome: Participants Who Achieved Response, Defined as Spironolactone Greater Than or Equal to 25 mg Daily
Description: The median percentages of participants who achieved a response are presented. Response means that the requirement was met. Non-response was indicated for subjects lost to follow-up, including death.
  The analysis was performed using a GEE model with a binomial family and a log link, a dependent variable of response per visit, fixed independent variables of randomised treatment, subject recruitment country, a per visit indicator variable and open-label period cohort. The common odds ratio was derived together with two-sided 95% confidence intervals.
Time Frame: From Month 1 (Visit 9) to Month 6 (Visit 14), up to 6 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 102 | 101
Percentage of participants | 81.4 | 49.5
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p < 0.001, GEE model; Odds Ratio (OR) = 4.33, 95% CI 2-sided [2.50 to 7.52] — An odds ratio greater than 1 indicated increased odds of response on SZC compared to placebo

4. Secondary Outcome: Time to First Hyperkalaemia (sK+ Greater Than 5.0mEq/L) Episode
Description: The time to first hyperkalaemia episode for participants on SZC compared to placebo during the randomised-withdrawal period, with hyperkalaemia defined as sK+ greater than 5.0 mEq/L as assessed by central laboratory, is presented in median time (days).
  The analysis was performed using a Cox regression model including randomised treatment group and subject recruitment country, adjusted for the stratification factor (hyperkalaemia vs normokalaemia at study entry). Placebo group used as reference level in Cox model.
Time Frame: From randomisation to the end of treatment (EOT) visit, up to 6 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 102 | 101
Days | 65.0 [35.00 to 98.00] | 9.0 [8.00 to 13.00]
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI [0.37 to 0.71] — A hazard ratio less than 1 favors SZC to be associated with a longer time to first hyperkalaemia episode than placebo

5. Secondary Outcome: Time to First Instance of Decrease or Discontinuation of Spironolactone Dose Due to Hyperkalaemia
Description: The time to first instance of decrease or discontinuation of spironolactone dose due to hyperkalaemia is presented in median time (days).
  The analysis was performed using a Cox regression model, adjusted for the stratification factor (hyperkalaemia vs normokalaemia at study entry).
Time Frame: From randomisation to the EOT visit, up to 6 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 102 | 101
Days | NA [NA to NA] — Median time to first event could not be calculated due to the low number of events. | NA [NA to NA] — Median time to first event could not be calculated due to the low number of events.
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p = 0.006, Regression, Cox; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.17 to 0.73] — A hazard ratio less than 1 favored SZC to be associated with a longer time to first instance of a decrease of spironolactone dose due to hyperkalaemia than placebo

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) at EOT
Description: The KCCQ is a 23-item instrument measuring, from the patients' perspectives, their heart failure-related symptoms, physical and social limitations, self-efficacy, and health-related quality of life (QoL) over the prior 2 weeks. It was scored as follows: Physical Limitation (items 1a-f), Symptom Stability (item 2), Symptom Frequency (items 3, 5, 7, and 9), Symptom Burden (items 4, 6, and 8), Self Efficacy (items 10 and 11), QoL (items 12, 13, and 14), and Social Limitation (items 15a-d). Scores were calculated by summing the responses within each domain and by taking the average. Scale scores were transformed to a 0 to 100 range, with 0 implying the lowest level of functioning and 100 for the highest level of functioning. The CSS was calculated as the average of Physical Limitation Score and Total Symptom Score (TSS) and the TSS was calculated as the average of Symptom Frequency and Symptom Burden Scores.
  The change from randomisation in KCCQ-CSS is reported.
Time Frame: At EOT visit (approximately 6 months post-randomisation)
Population: Full Analysis Set: all participants with more than 50% of responses available at a visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 72 | 59
Score on a scale | 71.27 (2.57) | 72.27 (2.36)
Statistical Analysis 1: Comparison: Randomized-withdrawal Phase - SZC Group vs Randomized-withdrawal Phase - Placebo Group; Test type: Superiority; p = 0.724, t-test, 2 sided; Least-squares Mean Difference = -1.01, 95% CI 2-sided [-6.64 to 4.63], Standard Error of Mean 2.84 — A least-squares mean difference greater than 0 favors SZC compared to placebo

7. Other Pre Specified Outcome: Location and Severity of Peripheral Oedema
Description: The location and severity of peripheral oedema that occurred during the randomised-withdrawal phase are presented. Participants with multiple peripheral oedema events were counted only once. The location of oedema is not mutually exclusive so multiple locations may apply for each participant.
Time Frame: During the randomised-withdrawal period and up to 14 days after discontinuation of SZC or placebo, up to 6.5 months
Population: Safety Set Randomised
Measure: Number; unit: Participants
Arm/Group | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
Number analyzed (Participants) | 22 | 16
Participants
  Location of oedema: pedal oedema | 13 | 10
  Location of oedema: ankle oedema | 17 | 13
  Location of oedema: pretibial oedema | 11 | 5
  Location of oedema: thigh oedema | 1 | 0
  Severity of pedal oedema - right side: trace | 4 | 3
  Severity of pedal oedema - right side: mild | 1 | 5
  Severity of pedal oedema - right side: moderate | 7 | 1
  Severity of pedal oedema - right side: severe | 0 | 0
  Severity of pedal oedema - left side: trace | 4 | 5
  Severity of pedal oedema - left side: mild | 2 | 4
  Severity of pedal oedema - left side: moderate | 7 | 1
  Severity of pedal oedema - left side: severe | 0 | 0
  Severity of ankle oedema - right side: trace | 4 | 4
  Severity of ankle oedema - right side: mild | 5 | 6
  Severity of ankle oedema - right side: moderate | 7 | 1
  Severity of ankle oedema - right side: severe | 0 | 0
  Severity of ankle oedema - left side: trace | 4 | 6
  Severity of ankle oedema - left side: mild | 5 | 6
  Severity of ankle oedema - left side: moderate | 8 | 1
  Severity of ankle oedema - left side: severe | 0 | 0
  Severity of pretibial edema - right side: trace | 2 | 1
  Severity of pretibial edema - right side: mild | 4 | 2
  Severity of pretibial edema - right side: moderate | 5 | 1
  Severity of pretibial edema - right side: severe | 0 | 0
  Severity of pretibial edema - left side: trace | 1 | 2
  Severity of pretibial edema - left side: mild | 3 | 2
  Severity of pretibial edema - left side: moderate | 7 | 1
  Severity of pretibial edema - left side: severe | 0 | 0
  Severity of thigh edema - right side: trace | 0 | 0
  Severity of thigh edema - right side: mild | 0 | 0
  Severity of thigh edema - right side: moderate | 1 | 0
  Severity of thigh edema - right side: severe | 0 | 0
  Severity of thigh edema - left side: trace | 0 | 0
  Severity of thigh edema - left side: mild | 0 | 0
  Severity of thigh edema - left side: moderate | 1 | 0
  Severity of thigh edema - left side: severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Open-label Run-in Phase (OLP): includes treatment-emergent adverse events (TEAEs) that occurred during the OLP and all AEs which occurred prior to first dose of SZC which worsen in severity following dosing during the OLP, up to 4-6 weeks Randomised-withdrawal Phase (RWP): includes TEAEs that occurred during the RWP and up to 14 days after discontinuation of SZC/placebo and all AEs which occurred prior to first dose which worsen in severity following dosing during the RWP, up to 6.5 months
Description: The AEs that occurred during the OLP and RWP are reported. The SZC group and Placebo group represent participants assessed during the RWP.
  OLP: Of the 366 participants who enrolled, 4 participants did not receive treatment and were excluded from the analysis.
  RWP: Of the 203 participants randomized (102 in the SZC group and 101 in the Placebo group), 1 participant from the SZC group did not receive treatment and was excluded from the analysis.
Groups:
- Open-label Run-in Phase: Participants with symptomatic heart failure with reduced ejection fraction who were taking no or low-dose spironolactone or eplerenone (<25 mg daily) at screening were enrolled and allocated to Cohort 1 (hyperkalaemic at study entry) or Cohort 2 (normokalaemic at study entry).
Arm/Group | Open-label Run-in Phase | Randomized-withdrawal Phase - SZC Group | Randomized-withdrawal Phase - Placebo Group
All-Cause Mortality (participants affected / at risk) | 7/362 | 2/101 | 2/101
Serious Adverse Events (participants affected / at risk) | 11/362 | 23/101 | 22/101
Other Adverse Events (participants affected / at risk) | 9/362 | 20/101 | 25/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Run-in Phase (N=362) | Randomized-withdrawal Phase - SZC Group (N=101) | Randomized-withdrawal Phase - Placebo Group (N=101)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (4) | 12 (14) | 4 (4)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Run-in Phase (N=362) | Randomized-withdrawal Phase - SZC Group (N=101) | Randomized-withdrawal Phase - Placebo Group (N=101)
Oedema peripheral (General disorders) | 3 (3) | 6 (6) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (9) | 12 (16) | 23 (34)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04676646/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04676646/SAP_001.pdf